CLINICAL TRIAL: NCT00554086
Title: Phase 2 Trial of Maximum Androgen Blockade (MAB) Dose Escalation From 50 mg to 150 mg Bicalutamide (Casodex) for Biochemical Failure in Prostate Cancer Patients
Brief Title: Open Label,Phase II Trial of MAB Dose Escalation OF Bicalutamide For Biochemical Failure In Prostate Cancer Patients.
Acronym: CHICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Laurence Klotz, Canadian Urology Research Consortium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6876L00008; NCT00260455 (obsolete NCT alias)
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escalating dose of Casodex from 50mg daily to 150 mg daily — Casodex dosage increase from 50mg to 150mg daily until baseline serum PSA is reduced by 50%

SUMMARY:
Multi-centre one year trial for patients who have rising PSA while on Casodex 50mg daily dose. Casodex dosage escalated to 150 mg tablet daily. Treatment will be continued until patient demonstrates clinical benefit at one year, PSA progression, toxicity, or withdrawal. Treatment will be continued after one year if patient demonstrates continued clinical benefit.

DETAILED DESCRIPTION:
The study will be a national, multicentre, open-label, phase II trial. Patients who have a rising PSA on MAB with bicalutamide 50 mg daily will be dose escalated to MAB with 150 mg bicalutamide daily. Subjects will receive trial treatment for 12 months, or until disease progression, unacceptable toxicity or withdrawal of consent. Open label treatment will be offered thereafter if the subject demonstrates clinical benefit at the end of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Men, over 18 years of age, with histologically-confirmed prostate cancer
3. Treatment with Zoladex (goserelin acetate) for greater than 3 months prior to Day 1
4. Serum testosterone level < 50 ng/ml
5. Current treatment with bicalutamide 50 mg daily.**
6. Two consecutive rises in PSA above a nadir value, with the absolute value of the latest PSA > 2.0 ng/ml.
7. Highest PSA level no greater than or equal to 30 ng/ml.
8. Life expectancy of greater than 1 year -

Exclusion Criteria:

1. Patients may not have received prolonged anti-androgen therapy other than with bicalutamide. Patients who have received short term (2 months or less) non-steroidal anti-androgen therapy with an agent other than bicalutamide to block flare are not excluded.*
2. PSA level greater than 30 ng/ml.
3. In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease which would make it undesirable for the patient to participate in the trial.
4. Subjects who have received prior chemotherapy.
5. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or superficial transitional cell carcinoma of the bladder.
6. Absolute neutrophil count less than 1.5 x 109/L or platelets less than 100 x 109/L.
7. Serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR).
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULRR.
9. Serum creatinine greater than 1.5 times -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-11; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Doubling of PSA | one year

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, Principal Investigator — Canadian Urology Research Consortium
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada